CLINICAL TRIAL: NCT02189837
Title: Double-blind, Randomized, Placebo-controlled, Single Site Study to Evaluate the Effects of Evolocumab (AMG 145) Treatment, Alone and in Combination With Atorvastatin, on Lipoprotein Kinetics
Brief Title: Effects on Lipoprotein Metabolism From PCSK9 Inhibition Utilizing a Monoclonal Antibody
Acronym: FLOREY
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20130194; FLOREY (Other: Amgen)
Record Dates: First submitted 2014-07-08; First posted 2014-07-15 (Estimated); Results first posted 2016-08-31 (Estimated); Last update posted 2018-10-03 (Actual); Status verified 2018-09

CONDITIONS: Primary Hyperlipidemia and Mixed Dyslipidemia
Keywords: Raised cholesterol; Cholesterol; Elevated Cholesterol; Hyperlipidemias; Dyslipidemias; Lipid Metabolism Disorders; Metabolic Diseases
MeSH Terms: conditions — Hypercholesterolemia; Hyperlipidemias; Dyslipidemias; Lipid Metabolism Disorders; Metabolic Diseases | interventions — evolocumab; Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo (Placebo Comparator): Participants received placebo subcutaneous injection once every 2 weeks on days 1, 15, 29 and 43 and placebo tablets once a day for up to 8 weeks.
  Interventions: Drug: Placebo to Evolocumab; Drug: Placebo to Atorvastatin
- Atorvastatin (Active Comparator): Participants received placebo subcutaneous injection once every 2 weeks on days 1, 15, 29 and 43 and 80 mg atorvastatin orally once a day for up to 8 weeks.
  Interventions: Drug: Atorvastatin; Drug: Placebo to Evolocumab
- Evolocumab (Experimental): Participants received 420 mg evolocumab by subcutaneous injection once every 2 weeks on days 1, 15, 29 and 43 and placebo tablets once a day for up to 8 weeks.
  Interventions: Biological: Evolocumab; Drug: Placebo to Atorvastatin
- Evolocumab and Atorvastatin (Experimental): Participants received 420 mg evolocumab by subcutaneous injection once every 2 weeks on days 1, 15, 29 and 43 and 80 mg atorvastatin orally once a day for up to 8 weeks.
  Interventions: Biological: Evolocumab; Drug: Atorvastatin

INTERVENTIONS:
Biological: Evolocumab — Administered by subcutaneous injection
  Other Names: AMG 145; Repatha
  Arms: Evolocumab; Evolocumab and Atorvastatin
Drug: Atorvastatin — Administered by mouth
  Other Names: LIPITOR®
  Arms: Atorvastatin; Evolocumab and Atorvastatin
Drug: Placebo to Evolocumab — Administered by subcutaneous injection
  Arms: Atorvastatin; Placebo
Drug: Placebo to Atorvastatin — Administered by mouth
  Arms: Evolocumab; Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled trial to evaluate the effect of evolocumab, atorvastatin, and combination therapy on lipoprotein kinetics.

ELIGIBILITY:
Inclusion Criteria:

* Fasting LDL-C at screening ≥ 100 mg/dL and ≤ 190 mg/dL
* Fasting triglycerides ≤ 150 mg/dL
* Body mass index (BMI) between 18.0 and 32.0 kg/m^2
* Framingham cardiac risk score 10% or less

Exclusion Criteria:

* Treatment with a lipid-regulating drug or over the counter supplement in the last 3 months prior to screening
* History of coronary heart disease (CHD) or CHD equivalent
* Uncontrolled hypertension
* Diabetes mellitus

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2014-07-08 (Actual); Primary Completion 2015-02-13 (Actual); Study Completion 2015-03-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (2):
- Australia (2):
  - Research Site, Adelaide, South Australia
  - Research Site, Nedlands, Western Australia

REFERENCES:
- [Background] Watts GF, Chan DC, Dent R, Somaratne R, Wasserman SM, Scott R, Burrows S, R Barrett PH. Factorial Effects of Evolocumab and Atorvastatin on Lipoprotein Metabolism. Circulation. 2017 Jan 24;135(4):338-351. doi: 10.1161/CIRCULATIONAHA.116.025080. Epub 2016 Dec 9. PMID 27941065
- [Background] Watts GF, Chan DC, Somaratne R, Wasserman SM, Scott R, Marcovina SM, Barrett PHR. Controlled study of the effect of proprotein convertase subtilisin-kexin type 9 inhibition with evolocumab on lipoprotein(a) particle kinetics. Eur Heart J. 2018 Jul 14;39(27):2577-2585. doi: 10.1093/eurheartj/ehy122. PMID 29566128
- [Background] Chan DC, Watts GF, Somaratne R, Wasserman SM, Scott R, Barrett PHR. Comparative Effects of PCSK9 (Proprotein Convertase Subtilisin/Kexin Type 9) Inhibition and Statins on Postprandial Triglyceride-Rich Lipoprotein Metabolism. Arterioscler Thromb Vasc Biol. 2018 Jul;38(7):1644-1655. doi: 10.1161/ATVBAHA.118.310882. Epub 2018 Jun 7. PMID 29880491
- [Derived] Chan DC, Watts GF, Coll B, Wasserman SM, Marcovina SM, Barrett PHR. Lipoprotein(a) Particle Production as a Determinant of Plasma Lipoprotein(a) Concentration Across Varying Apolipoprotein(a) Isoform Sizes and Background Cholesterol-Lowering Therapy. J Am Heart Assoc. 2019 Apr 2;8(7):e011781. doi: 10.1161/JAHA.118.011781. PMID 30897995
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 2 centers in Australia. The first participant was enrolled on 08 July 2014, and the last participant enrolled on 15 December 2014.
Pre-assignment Details: Participants who met eligibility criteria underwent an initial 4 week run-in period of dietary stabilization before randomization. Randomization was stratified based on screening low-density lipoprotein (LDL-C) concentration (< 130 mg/dL vs ≥ 130 mg/dL)
Period: Overall Study
Arm/Group | Placebo | Atorvastatin | Evolocumab | Evolocumab and Atorvastatin
Started | 22 | 23 | 23 | 21
Received Treatment | 21 | 22 | 22 | 20
Completed | 20 | 22 | 20 | 19
Not Completed | 2 | 1 | 3 | 2
Not completed — Withdrawal by Subject | 2 | 1 | 3 | 1
Not completed — Sponsor Decision | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The full analysis set includes all randomized participants who received any study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Atorvastatin | Evolocumab | Evolocumab and Atorvastatin | Total
Number analyzed (Participants) | 21 | 22 | 22 | 20 | 85
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.9 (12.7) | 30.4 (7.4) | 33.5 (11.6) | 31.0 (9.8) | 32.2 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 21 | 22 | 22 | 20 | 85
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 2 | 1 | 3 | 7
  Black or African American | 0 | 0 | 0 | 3 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  White | 19 | 20 | 20 | 14 | 73
  Other | 1 | 0 | 1 | 0 | 2
  Mixed Race | 0 | 0 | 0 | 0 | 0
Screening LDL-C Level [Number; unit: participants]
  < 130 mg/dL | 9 | 9 | 9 | 8 | 35
  ≥ 130 mg/dL | 12 | 13 | 13 | 12 | 50
LDL-C Concentration [Mean (Standard Deviation); unit: mg/dL] — LDL-C was measured using ultracentrifugation
  mg/dL | 118.1 (18.1) | 123.2 (21.3) | 118.2 (18.4) | 116.5 (23.7) | 119.1 (20.2)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Low-density Lipoprotein (LDL) Apolipoprotein B-100 Fractional Catabolic Rate (FCR)
Description: The fractional catabolic rate (the percentage of apolipoprotein B-100 in LDL which is replaced, transferred or lost per unit of time) was measured at Baseline and Day 50 over 5 consecutive days using the stable isotope tracer, D3-leucine. LDL particles were isolated from plasma by sequential ultracentrifugation, and isotopic enrichment was determined using gas chromatography-mass spectrometry. Mathematical modelling of the protein enrichment data was used to estimate protein catabolism.
Time Frame: Baseline (5 days prior to Day 1) and Day 50; plasma samples for fasting lipids were obtained at 0, 5, 10, 20, 30, 40, and 60 min, as well as at 1.5, 2, 2.5, 3, 4, 5, 6, 8, and 10 hours, and 2, 3, 4 and 5 days after D3-leucine administration.
Population: Efficacy Analysis Set including all randomized and dosed participants who completed baseline and Day 50 measurements.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Atorvastatin | Evolocumab | Evolocumab and Atorvastatin
Number analyzed (Participants) | 20 | 22 | 20 | 19
percent change | -5.07 (26.06) | 74.13 (24.84) | 83.70 (26.06) | 310.48 (26.68)
Statistical Analysis 1: Comparison: Placebo vs Evolocumab; The superiority of evolocumab monotherapy to placebo was tested using a 2-sided p-value at a significance level of 0.05; Test type: Superiority or Other; p = 0.018, ANCOVA; Model includes terms for the 2 factors in the factorial design (placebo or evolocumab and oral placebo or statin), their interaction, and LDL-C level; LS Mean Treatment Difference = 88.76, 95% CI 2-sided [15.73 to 161.80], Standard Error of Mean 36.67
Statistical Analysis 2: Comparison: Atorvastatin vs Evolocumab and Atorvastatin; The treatment effect of evolocumab plus atorvastatin compared with placebo plus atorvastatin was estimated and a nominal p-value is provided; Test type: Superiority or Other; p < 0.001, ANCOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = 236.35, 95% CI 2-sided [164.02 to 308.69], Standard Error of Mean 36.32
Statistical Analysis 3: Comparison: Placebo vs Atorvastatin vs Evolocumab vs Evolocumab and Atorvastatin; To assess whether the treatment effect of evolocumab compared with placebo depended on being administered alone or combined with atorvastatin, the interaction was tested, i.e., the difference between the treatment difference versus the respective placebo group for the evolocumab+atorvastatin group and the evolocumab group was calculated; Test type: Superiority or Other; p = 0.005, ANCOVA; [statistical method as in outcome 1, analysis 1]; Treatment Effect = 147.59, 95% CI 2-sided [44.80 to 250.38], Standard Error of Mean 51.61

2. Secondary Outcome: Percent Change From Baseline in LDL-C at Day 50
Description: LDL-C was measured using ultrcentrifugation.
Time Frame: Baseline and Day 50
Population: Efficacy Analysis Set with available data at both time points
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Atorvastatin | Evolocumab | Evolocumab and Atorvastatin
Number analyzed (Participants) | 19 | 22 | 18 | 17
percent change | -0.65 (3.09) | -45.25 (2.86) | -57.79 (3.15) | -83.19 (3.24)
Statistical Analysis 1: Comparison: Placebo vs Evolocumab; Test type: Superiority or Other; p < 0.001, ANCOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -57.14, 95% CI [-65.91 to -48.38], Standard Error of Mean 4.40
Statistical Analysis 2: Comparison: Atorvastatin vs Evolocumab and Atorvastatin; Test type: Superiority or Other; p < 0.001, ANCOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -37.95, 95% CI 2-sided [-46.55 to -29.34], Standard Error of Mean 4.31
Statistical Analysis 3: Comparison: Placebo vs Atorvastatin vs Evolocumab vs Evolocumab and Atorvastatin; Test type: Superiority or Other; p = 0.003, ANCOVA; [statistical method as in outcome 1, analysis 1]; Treatment Effect = 19.20, 95% CI 2-sided [6.93 to 31.47], Standard Error of Mean 6.15

3. Secondary Outcome: Percent Change From Baseline in LDL Apolipoprotein B-100 Production Rate (PR)
Description: The production rate of apolipoprotein B-100 in LDL was measured at Baseline and Day 50 over 5 consecutive days using the stable isotope tracer, D3-leucine. LDL particles were isolated from plasma by sequential ultracentrifugation and isotopic enrichment was determined using gas chromatography-mass spectrometry. Mathematical modelling of the protein enrichment data was used to estimate the production rate.
Time Frame: Baseline and Day 50
Population: Efficacy Analysis Set
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Atorvastatin | Evolocumab | Evolocumab and Atorvastatin
Number analyzed (Participants) | 20 | 22 | 20 | 19
percent change | -3.80 (7.40) | -3.27 (7.05) | -20.45 (7.40) | -35.93 (7.57)
Statistical Analysis 1: Comparison: Placebo vs Evolocumab; Test type: Superiority or Other; p = 0.11, ANCOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -16.65, 95% CI 2-sided [-37.37 to 4.08], Standard Error of Mean 10.41
Statistical Analysis 2: Comparison: Atorvastatin vs Evolocumab and Atorvastatin; Test type: Superiority or Other; p = 0.002, ANCOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -32.66, 95% CI 2-sided [-53.19 to -12.13], Standard Error of Mean 10.31
Statistical Analysis 3: Comparison: Placebo vs Atorvastatin vs Evolocumab vs Evolocumab and Atorvastatin; Test type: Superiority or Other; p = 0.28, ANCOVA; [statistical method as in outcome 1, analysis 1]; Treatment Effect = -16.01, 95% CI 2-sided [-45.18 to 13.16], Standard Error of Mean 14.65

4. Secondary Outcome: Percent Change From Baseline in Lipoprotein (a) Fractional Catabolic Rate (FCR)
Description: The fractional catabolic rate (the percentage of lipoprotein(a) (Lp[a]) which is replaced, transferred or lost per unit of time) was measured at Baseline and Day 50 over 5 consecutive days using the stable isotope tracer, D3-leucine. Lp(a) was isolated from plasma using an immunoprecipitation method employing immunomagnetic beads and polyacrylamide gel electrophoresis. Isotopic enrichment was determined using gas chromatography-mass spectrometry. Mathematical modelling of the protein enrichment data was used to estimate protein catabolism.
Time Frame: as for outcome 1
Population: Efficacy Analysis Set with available data
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Atorvastatin | Evolocumab | Evolocumab and Atorvastatin
Number analyzed (Participants) | 16 | 17 | 14 | 16
percent change | 7.49 (9.17) | 25.52 (8.92) | 5.37 (9.81) | 64.57 (9.23)
Statistical Analysis 1: Comparison: Placebo vs Evolocumab; The superiority of evolocumab monotherapy to placebo was tested using a 2-sided p-value at a significance level of 0.05; Test type: Superiority or Other; p = 0.87, ANCOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -2.12, 95% CI 2-sided [-28.94 to 24.70], Standard Error of Mean 13.40
Statistical Analysis 2: Comparison: Atorvastatin vs Evolocumab and Atorvastatin; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.003, ANCOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = 39.06, 95% CI 2-sided [13.52 to 64.59], Standard Error of Mean 12.76
Statistical Analysis 3: Comparison: Placebo vs Atorvastatin vs Evolocumab vs Evolocumab and Atorvastatin; [analysis description as in outcome 1, analysis 3]; Test type: Superiority or Other; p = 0.030, ANCOVA; [statistical method as in outcome 1, analysis 1]; Treatment Effect = 41.18, 95% CI 2-sided [4.15 to 78.20], Standard Error of Mean 18.50

5. Secondary Outcome: Percent Change From Baseline in Lipoprotein(a) Production Rate (PR)
Description: The production rate of lipoprotein(a) was measured at Baseline and Day 50 over 5 consecutive days using the stable isotope tracer, D3-leucine. Lp(a) was isolated from plasma using an immunoprecipitation method employing immunomagnetic beads and polyacrylamide gel electrophoresis. Isotopic enrichment was determined using gas chromatography-mass spectrometry. Mathematical modelling of the protein enrichment data was used to estimate protein catabolism.
Time Frame: Baseline and Day 50
Population: Efficacy Analysis Set with available data
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Atorvastatin | Evolocumab | Evolocumab and Atorvastatin
Number analyzed (Participants) | 16 | 17 | 14 | 16
percent change | 3.52 (7.94) | -6.88 (7.72) | -35.91 (8.49) | 16.40 (7.99)
Statistical Analysis 1: Comparison: Placebo vs Evolocumab; Test type: Superiority or Other; p = 0.001, ANCOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -39.43, 95% CI 2-sided [-62.66 to -16.21], Standard Error of Mean 11.60
Statistical Analysis 2: Comparison: Atorvastatin vs Evolocumab and Atorvastatin; Test type: Superiority or Other; p = 0.039, ANCOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = 23.28, 95% CI 2-sided [1.16 to 45.40], Standard Error of Mean 11.05
Statistical Analysis 3: Comparison: Placebo vs Atorvastatin vs Evolocumab vs Evolocumab and Atorvastatin; Test type: Superiority or Other; p < 0.001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Treatment Effect = 62.72, 95% CI 2-sided [30.65 to 94.79], Standard Error of Mean 16.02

ADVERSE EVENTS:
Time Frame: From first dose of study drug until day 73
Description: Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
Arm/Group | Placebo | Atorvastatin | Evolocumab | Evolocumab and Atorvastatin
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/22 | 0/22 | 1/20
Other Adverse Events (participants affected / at risk) | 5/21 | 12/22 | 14/22 | 10/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=21) | Atorvastatin (N=22) | Evolocumab (N=22) | Evolocumab and Atorvastatin (N=20)
Liver injury (Hepatobiliary disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=21) | Atorvastatin (N=22) | Evolocumab (N=22) | Evolocumab and Atorvastatin (N=20)
Abdominal pain (Gastrointestinal disorders) | 0 | 2 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 3 | 2 | 2
Influenza like illness (General disorders) | 0 | 0 | 2 | 0
Nasopharyngitis (Infections and infestations) | 1 | 1 | 2 | 0
Pharyngitis (Infections and infestations) | 0 | 2 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 2 | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 0 | 2 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1 | 0
Headache (Nervous system disorders) | 2 | 5 | 8 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.